CLINICAL TRIAL: NCT01836133
Title: Efficacy and Safety of Erlotinib (Tarceva® ) Therapy in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) , Subtype Adenocarcinoma, Who Have Good Performance Status (PS 0-1) - ELEMENT
Brief Title: An Observational Study of Tarceva (Erlotinib) in Participants With Locally Advanced or Metastatic Adenocarcinoma Non-Small Cell Lung Cancer (ELEMENT)
Acronym: ELEMENT
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28282
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Erlotinib 150 mg: Participants received 150 mg erlotinib once daily, orally, as tablets, until disease progression or unacceptable toxicity, up to 3 years.
  Interventions: Drug: Erlotinib 150 mg

INTERVENTIONS:
Drug: Erlotinib 150 mg

SUMMARY:
This multicenter, observational study will evaluate the efficacy and safety of Tarceva (erlotinib) in participants with locally advanced or metastatic adenocarcinoma non-small cell lung cancer and an ECOG performance status of 0-1. Eligible participants receiving Tarceva according to the Summary of Product Characteristics and local label will be followed for the duration of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Histologically or cytologically confirmed, locally advanced (Stage IIIb) or metastatic (Stage IV) adenocarcinoma non-small cell lung cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematologic, renal and liver function
* Participant initiating treatment with Tarceva according to the Summary of Product Characteristics

Exclusion Criteria:

* Any contraindications to treatment with Tarceva according to the Summary of Product Characteristics and local label
* Any other malignancies within the previous 5 years, except for in situ carcinoma of the cervix and basal and squamous cell carcinoma of the skin
* Previous systemic anti-cancer treatment with HER1/EGFR inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with locally advanced or metastatic adenocarcinoma non-small cell lung cancer, with ECOG performance status of 0-1
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Serbia (5):
  - Clinical Center of Serbia; Institute For Pulmology, Belgrade
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Military Medical Academy; Clinic for Pulmonology, Belgrade
  - Institute for pulmonary diseases of Vojvodina, Kamenitz
  - Clinical Center Nis; Clinic for pulmonary diseases Knez Selo, Knez-Selo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib 150 mg
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from initial dose of erlotinib to progression or death from any cause.
Time Frame: Approximately 3 years
Population: The effectiveness analysis population included all enrolled participants in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 70
months | 2.7 [2.4 to 3.0]

2. Secondary Outcome: Percentage of Participants With Overall Response
Description: Overall response was defined, based on response evaluation criteria in solid tumours (RECIST) v 1.1, as complete response (CR) plus partial response (PR). CR: complete disappearance of all target lesions; PR: at least 30% decrease in the sum of the longest diameter of all target lesions taking as reference the baseline sum of all target lesions.
Time Frame: Approximately 3 years
Population: The effectiveness analysis population included all enrolled participants in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 70
Percentage of participants | 8.57 [3.67 to 17.78]

3. Secondary Outcome: Proportions of Participants With Adverse Events (AEs), Serious AEs, and AEs of Special Interest (AESIs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant, according to national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) criteria version 4.0. An AESI was defined as interstitial pulmonary disease.
Time Frame: Baseline up to 3 years
Population: The safety analysis population included all enrolled participants who received a single dose of erlotinib.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Erlotinib 150 mg
Number analyzed (Participants) | 70
Proportion of participants
  AEs | 0.56 [0.44 to 0.67]
  SAEs | 0.27 [0.18 to 0.39]
  AESIs | 0 [NA to NA] — 95% Confidence Interval was not calculated because no AESIs were reported.

ADVERSE EVENTS:
Time Frame: Baseline up to 3 years
Description: All enrolled participants were included in the safety population.
Arm/Group | Erlotinib 150 mg
Serious Adverse Events (participants affected / at risk) | 19/70
Other Adverse Events (participants affected / at risk) | 21/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg (N=70)
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 2
Pyrexia (General disorders) | 1
Fatigue (General disorders) | 1
Disease progression (General disorders) | 2
Sudden death (General disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 2
Pneumonia (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Conjuctivitis (Infections and infestations) | 1
Weight decreased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Azotaemia (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib 150 mg (N=70)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Paronychia (Infections and infestations) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.